CLINICAL TRIAL: NCT02271789
Title: Low-cost, Noninvasive Method to Assess Pulpal Vitality
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial study
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Petra Wilder-Smith, DDS., PhD., Professor, Director of Dentistry, University of California, Irvine
Other Study IDs: 20141390
Record Dates: First submitted 2014-10-09; First posted 2014-10-22 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Other Dental Disease/Condition of Teeth/Supporting Structure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: problematic tooth — problematic tooth

SUMMARY:
The purpose of this research study is to find a new way of using light to measure the blood flow within the tooth.

The researcher develop dental Laser Speckle imaging system tool that can use for exam condition of the tooth. This device is reliable method to provide information to dentists and endodontists during oral examination.

DETAILED DESCRIPTION:
In additional to routine oral exam the researcher can use the Laser Speckle imaging system probe with low-level light shine to the problematic tooth to collect blood flow information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 30.
* Have one or more teeth requiring endodontic treatment.

Exclusion Criteria:

* Participation in other study within 3 months of enrollment in this study,
* Pregnant Women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from affiliated researcher at Dentists clinic in Orange Country and will be referred to investigator at University of California Irvine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Healthy tooth | up to 4 weeks
  Healthy tooth

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS., PhD, Principal Investigator — Beckman Laser Instiute, UCI
Locations (1):
- Beckman Laser Institute, UCI, Irvine, California, United States